CLINICAL TRIAL: NCT04677751
Title: Clinical and Electrographic Changes in RNS System Patients with Acupuncture Treatment
Brief Title: Clinical and Electrographic Changes in Responsive Neurostimulation System (RNS) Patients with Acupuncture Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Olga Rodziyevska, Physician Assistant, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HSC-MS-20-0743
Record Dates: First submitted 2020-12-15; First posted 2020-12-21 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-07

CONDITIONS: Epilepsy
Keywords: acupuncture; RNS; seizure
MeSH Terms: conditions — Epilepsy; Seizures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Experimental group (Experimental)
  Interventions: Device: Acupuncture intervention

INTERVENTIONS:
Device: Acupuncture intervention — Participants will undergo 12 weeks of acupuncture therapy. There will be one 40 minute-1 hour. session per week.

SUMMARY:
The purpose of this study is to determine effects of Acupuncture on a Patient's mood and cognition,evaluate changes in clinically-reported seizure frequency and severity and analyze effects of Acupuncture on electrographic epileptiform activity stored by the RNS System

ELIGIBILITY:
Inclusion Criteria:

* Patient implanted with the RNS system
* Patient can undergo 12 weeks of acupuncture
* Patient is able remain on stable medications for 12 weeks
* Patient is able to remain on stable Detection and Stimulation settings for 12 weeks
* Patient or/and caregiver is able to understand and sign informed consent and HIPAA authorization
* Patient or caregiver able to maintain a seizure diary for duration of study

Exclusion Criteria:

* Patient and /or caregiver is unable to sign informed consent to study
* Patient has a bleeding disorder, pacemaker, or pregnant

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Percent change in number of disabling clinical seizures | Baseline,12 weeks post treatment
  This will be measured by self reporting journals
Changes in seizure severity | Baseline,12 weeks post treatment
  This will be measured by self reporting journals

SECONDARY OUTCOMES:
Change in cognition and mood as assessed by the Quality Of Life In Epilepsy (QOLIE-10) questionnaire | Baseline,12 weeks post treatment
  This is a 10 item questionnaire. Score ranges from 1-6,a higher number indicating a worse outcome.
Change in cognition and mood as assessed by the Patient Health Questionnaire (PHQ-9) | Baseline,12 weeks post treatment
  PHQ-9 score can range from 0 to 27,each of the 9 items can be scored from 0 (not at all) to 3 (nearly every day).
Change in cognition and mood as assessed by the Generalized Anxiety Disorder 7-item (GAD-7) scale | Baseline,12 weeks post treatment
  This is a 7 item questionnaire. Each question is scored form 0(not at alll) to 3(nearly every day)
Average number of detections of seizures per-day (as stored by the RNS System) | Baseline
Average number of detections of seizures per-day (as stored by the RNS System) | end of 1 month
Average number of detections of seizures per-day (as stored by the RNS System) | end of 2 months
Average number of detections of seizures per-day (as stored by the RNS System) | end of 3 months
Average number of detections of seizures per-day (as stored by the RNS System) | 1 month after last treatment

CONTACTS AND LOCATIONS:
Overall Officials: Olga Rodziyevska, MS,PA-C, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No